CLINICAL TRIAL: NCT06037434
Title: A Prospective Controlled Study for the Treatment Effect of Different Intervention Strategies for Pediatric Mitral Regurgitation--A Multicenter Prospective Cohort Study of Innovative Drug Therapy for Pediatric Mitral Regurgitation
Brief Title: Study of Innovative Drug Treatment Therapy for Pediatric Mitral Regurgitation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Shanghai Children's Medical Center (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Guangzhou Women and Children's Medical Center (Other); Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Shoujun Li, Director of Congenital Heart Surgery Center, China National Center for Cardiovascular Diseases
Other Study IDs: 2022-GSP-GG-19-1
Record Dates: First submitted 2023-09-06; First posted 2023-09-14 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Congenital Mitral Insufficiency
Keywords: congenital heart disease; mitral regurgitation; drug therapy
MeSH Terms: conditions — Heart Defects, Congenital; Mitral Valve Insufficiency | interventions — Captopril; Metoprolol; Spironolactone; Torsemide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Modified Drug Therapy Group: Patient in this group will undergo a one-year course of medication, including Captopril(tablet, 0.3mg/kg, tid), Metoprolol(tablet, 0.2mg/kg, bid), Spironolactone(tablet, 2-4mg/kg, bid), Torsemide(tablet, 0.2-0.5mg/mg, bid), and Potassium Citrate(powder, 0.06g/kg, tid).
  Interventions: Drug: Captopril Tablets; Drug: Metoprolol Oral Tablet; Drug: Spironolactone Tablets; Drug: Torsemide Tablets; Drug: Potassium citrate powder
- the Traditional Drug Therapy Group: Patient in this group will undergo a one-year course of medication, including Torsemide(tablet, 0.2-0.5mg/mg, bid) and Potassium Citrate(powder, 0.06g/kg, tid).
  Interventions: Drug: Torsemide Tablets; Drug: Potassium citrate powder

INTERVENTIONS:
Drug: Captopril Tablets — 0.3mg/kg, tid
  Groups: Modified Drug Therapy Group
Drug: Metoprolol Oral Tablet — 0.2mg/kg, bid
  Groups: Modified Drug Therapy Group
Drug: Spironolactone Tablets — 2-4mg/kg, bid
  Groups: Modified Drug Therapy Group
Drug: Torsemide Tablets — 0.2-0.5mg/mg, bid
Drug: Potassium citrate powder — 0.06g/kg, tid

SUMMARY:
The goal of this observational study is to compare the safety and effectiveness of a modified drug therapy with traditional drug therapy in pediatric patients with mild to moderate mitral valve regurgitation.

The main questions it aims to answer are:

* Can a modified drug therapy improve both left ventricular and mitral valve function in pediatric patients with mild to moderate mitral valve regurgitation?
* Can the adverse drug reactions caused by the modified drug therapy be non-inferior (clinically acceptable) to those of the traditional drug therapy? Participants will be assigned to either the Modified Drug Therapy Group (comprising angiotensin-converting enzyme inhibitor (ACE-I), beta-blockers, diuretics, potassium supplements, and spironolactone) or the Traditional Drug Therapy Group (diuretics and potassium supplements) based on personal preferences and clinical assessments by their attending physicians. They will undergo a one-year course of medication. Additionally, echocardiography, electrocardiograms, complete blood counts, biochemical tests, and measurements of N-terminal pro-brain natriuretic peptide (NT-proBNP) were conducted before the initiation of medication therapy and at 3 months, 6 months, and 12 months after treatment commencement.

Researchers will compare the Modified Drug Therapy Group and the Traditional Drug Therapy Group to see if the recurrence rate of moderate to severe mitral valve regurgitation, as assessed by echocardiography after 12 months of treatment, is lower in the former than in the latter.

ELIGIBILITY:
Inclusion Criteria:

* < 14 years old
* had not undertake mitral valve surgery before
* moderate to severe mitral regurgitation

Exclusion Criteria:

* moderate to severe mitral regurgitation which concommitant with other cardiac malformation which can not be correct or can only perform palliative surgery
* concommitant with mitral stenosis
* ischemic mitral regurgitation (for example, concommitant with anomalous origin of coronary artery)
* Barlow syndrome
* dysplasia of mitral leaflet
* complete/Partial endocardial cushion defect
* common atrioventricular valve
* atrioventricular common channel
* cardiomyopathy
* other mitral valve surgery contraindications
* moderate to severe mitral regurgitation requires mitral valve surgery

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under the age of 14 with moderate to severe mitral valve regurgitation, without contraindications for mitral valve repair, and without an immediate need for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-08-09 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the recurrence rate of moderate to severe mitral valve regurgitation | after 12 months of treatment
  During follow-up visits, echocardiographic examination is conducted to measure the degree of mitral valve regurgitation. If it falls within the moderate to severe range, it is recorded as a recurrence.

SECONDARY OUTCOMES:
Improvement in symptoms | after 12 months of treatment
  Based on patient and caregiver descriptions, if symptoms such as chest discomfort, shortness of breath, and delayed development show improvement following physical activity, it is recorded as an improvement in symptoms.
Change in left ventricular ejection fraction | after 12 months of treatment
  Based on the echocardiogram, measurements are taken for left ventricular ejection fraction.
Change in left ventricular end-diastolic diameter | after 12 months of treatment
  Based on the echocardiogram, measurements are taken for left ventricular end-diastolic diameter.
NT-proBNP level | after 12 months of treatment
  The trend in NT-proBNP levels.
Incidence rate of drug adverse reactions | after 12 months of treatment
  The incidence of abnormalities in complete blood count, electrolytes, liver and kidney function, and cardiac enzymes.

CONTACTS AND LOCATIONS:
Overall Officials: Shoujun Li, MD, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No